CLINICAL TRIAL: NCT02827344
Title: Feasibility Study of PD-L1 Expression Analysis on Circulating Tumor Cells by Immunocytochemistry and MDSCs Level Evolution Analysis in Non-small Cell Lung Cancer Treated With PD-L1 or PD1 Inhibitor
Brief Title: PDL-1 Expression on Circulating Tumor Cells in Non-small Cell Lung Cancer
Acronym: IMMUNO-PREDICT
Status: Completed | Type: Observational
Sponsor: University Hospital, Toulouse (Other)
Responsible Party: Sponsor
Other Study IDs: 15 7737 02
Record Dates: First submitted 2016-07-06; First posted 2016-07-11 (Estimated); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: Lung Cancer
Keywords: PD-1/PD-L1; Immune checkpoints; Immunotherapy; lung cancer; circulating tumor cells; immunocytochemistry; ISET; MDSC; Stage IV non-small cell lung cancer
MeSH Terms: conditions — Lung Neoplasms; Neoplastic Cells, Circulating; Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — * Peripheral blood sample
  * Circulating tumor cells isolated from peripheral blood sample
  * MDSCs : immature myeloid cells that inhibit T cell functions rate analysis from peripheral blood sample
  * Tissue
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Stage IV non-small cell lung cancer: Intervention to be done are :
  - Blood sample collection for CTC and MDSC analysis
  Interventions: Biological: blood sample collection for CTC and MDSC analysis

INTERVENTIONS:
Biological: blood sample collection for CTC and MDSC analysis — * Isolation of circulating tumor cells from 2 tubes by ISET filtration module. Peripheral blood samples will be collected for CTC analysis within 7 days before commencing treatment (defined as baseline) and following four cycles of immunotherapy,
  * Analysis of PD-L1 and PD-L2 expression by immunocytochemistry on CTC
  * Analysis of the expression of PD-L1, PD-L2 , CTLA4 on the histological specimen by immunohistochemistry

SUMMARY:
Immunotherapy is probably, since the development of therapies targeting EGFR mutations or ALK rearrangement, the most attractive therapeutic perspective in the management of metastatic lung cancer. Among the compounds tested, the inhibitors of the immune checkpoint PROGRAMME DEATH 1 / PROGRAMME DEATH LIGAND 1 (PD-1/PD-L1) have been tested in numerous clinical trials with recently published positive results leading to the approval of one drug in the USA and an expanded access program for two drugs in France. PROGRAMME DEATH LIGAND 1 (PD-L1) expression by tumor cells is strongly associated with the response to such molecules so that the participation in various clinical trials is currently reserved for patients expressing this biomarker and therefore justifies a new invasive biopsy (bronchoscopic or CT-guided) representing a considerable drag on the access to these treatments. Circulating tumor cells (CTCs) isolated by Isolation by Size of Tumor Cells (ISET) offer a direct and non-invasive access to the tumor. It has already been demonstrated that molecular characterization (EGFR, ALK) on these blood samples is possible. We propose to demonstrate the feasibility of the analysis PDL-1 expression in these cells by immunocytochemistry.

Myeloid-Derived Suppressor Cells (MDSCs) are immature myeloid cells that inhibit T cell functions and thus promote tumor growth. These cells frequently express PD-L1. We propose to test whether MDSCs level and its evolution during treatment with PD1 inhibitor is correlated to the response to these drugs.

The main objective of this study is to demonstrate the feasibility of the analysis of PD-L1 expression on CTC

ELIGIBILITY:
Inclusion Criteria:

* Stage IV non-small cell lung cancer patient prior to start immunotherapy treatment
* Patients with World Health Organization (WHO) performance status 0-3
* Patients who were informed and had non opposition form signed by investigator
* Patients with healthcare insurance system affiliation

Exclusion Criteria:

* Prior malignancy within 5 years of study entry
* Refusal to participate
* Patient under legal protection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Stage IV non small lung cancer patients
Sampling Method: Non-Probability Sample
Enrollment: 216 (Actual)
Dates: Start 2015-10-01 (Actual); Primary Completion 2021-10 (Actual); Study Completion 2021-12 (Actual)

PRIMARY OUTCOMES:
Feasibility of analysis of PDL-1 expression on circulating tumor cells as assessed by immunocytochemistry analysis | Through the end of study (12 months)
  Prior to immunotherapy, after four cycle of immunotherapy

SECONDARY OUTCOMES:
Percentage of CTC expressing PD-L1 after four cycle of immunotherapy as assessed by immunocytochemistry analysis | Through the end of study (12 months)
  Prior to immunotherapy, after four cycle of immunotherapy
Evolution of MDSCs count in response to treatment as assessed by MDSCs analysis | Through the end of study (12 months)
  Prior to immunotherapy, after four cycle of immunotherapy

CONTACTS AND LOCATIONS:
Overall Officials: Nicolas GUIBERT, PH, Principal Investigator — University Hospital of Toulouse
Locations (1):
- Larrey Hospital, Toulouse, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Guibert N, Jones G, Beeler JF, Plagnol V, Morris C, Mourlanette J, Delaunay M, Keller L, Rouquette I, Favre G, Pradines A, Mazieres J. Targeted sequencing of plasma cell-free DNA to predict response to PD1 inhibitors in advanced non-small cell lung cancer. Lung Cancer. 2019 Nov;137:1-6. doi: 10.1016/j.lungcan.2019.09.005. Epub 2019 Sep 6. PMID 31518912
- [Result] Guibert N, Pradines A, Favre G, Mazieres J. [Finding mutations of interest in circulating tumor DNA helps predict immunotherapy response in lung cancer]. Med Sci (Paris). 2020 May;36(5):437-439. doi: 10.1051/medsci/2020068. Epub 2020 May 26. No abstract available. French. PMID 32452359